CLINICAL TRIAL: NCT01719510
Title: Study of the Digestive Colonization of the Newborn Children by the Streptococcus of the Group B
Brief Title: Interest of the Detection of Hyper-virulent Clone ST17 of Group B Strep (GBS) for the Prevention of Neonatal GBS Meningitis
Acronym: Col-Strepto B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: P111008
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Neonatal Infections Colonize With Group B Streptococci
Keywords: Group B Streptococcus,; Vaginal screening; Per partum antibiotic prophylaxis; Meningitis; Neonatal infection; PCR; Streptococcus agalactiae.
MeSH Terms: conditions — Meningitis | interventions — Sampling Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positive Group B Streptococcus vaginal sample (Other): At time of delivery we will performed vaginal swabs in two groups: women tested positive for GBS at 35-37 weeks and women with risk of neonatal infection.
  For all women included will be achieved in the delivery room:
  a blood sample to the mother and a sampling of umbilical cord blood. Newborns will have a search for GBS (standard culture) in the stools and the pharynx.
  For mothers, the collection of milk when breastfeeding.
  Interventions: Other: Samples

INTERVENTIONS:
Other: Samples — At time of delivery we will performed vaginal swabs in two groups: women tested positive for GBS at 35-37 weeks and women with risk of neonatal infection.
  For both groups:
  * one swab for GBS detection by real-time PCR
  * the second swab for GBS detection by conventional bacteriological techniques and sent to the bacteriology laboratory.
  For all women included will be achieved in the delivery room:
  1. To the mother: A blood sample of 5 ml at the time of the implementation of the IV line.
  2. A sampling of umbilical cord blood.
  Newborns of mothers included (group 1 and 2) will have a search for GBS (standard culture) in the stools and the pharynx prior to return home.
  For mothers, the collection of 3-5 ml of milk when breastfeeding.

SUMMARY:
The main objective of this study : Demonstrate that GBS (group B streptococci) "ST-17" colonize and persist to 60 days twice in the digestive tract of newborns that strains of GBS non-ST-17.

Secondary objectives:Determine:

* The frequency of colonization with GBS ST-17 and GBS non-ST-17 of at risk pregnant women.
* The frequency of colonization of neonates by GBS ST-17 at birth.
* The preferential site of colonization in the mother (rectum, vagina, breast milk).
* The kinetics of colonization after birth in the newborn.
* The sensitivity and specificity of different GBS detection methods (conventional phenotypic versus molecular) in the different types of samples from the mother and the newborn.

DETAILED DESCRIPTION:
Women tested positive for GBS during systematic vaginal screening at 35-37 weeks, will be proposed to participate to the study and will be included after reading the information letter and signature the consent form.

INCLUSION (D0 at time of delivery)

In the labor ward, two women's groups 1 and 2:

Group 1 = Women tested positive for GBS pre-selected and included in the protocol (see pre-inclusion) Group 2 = Women without antenatal vaginal screening and at risk of neonatal infection.

For both groups, at time of delivery:

At the beginning of the labour performed vaginal swabs (PV0):

* one swab for GBS detection by real-time PCR using the Cepheid technique conducted in the labor ward by the midwife.
* the second swab for GBS detection by conventional bacteriological techniques and sent to the bacteriology laboratory.

For all women included (Group 1 and Group 2 women with a positive GBS vaginal sample) will be achieved in the delivery room:

1. To the mother: A blood sample of 5 ml at the time of the implementation of the IV line.
2. A sampling of umbilical cord blood. Newborns of mothers included (group 1 and 2) will have a search for GBS (standard culture) in the stools and the pharynx prior to return home. Samples will be sent to the bacteriology laboratory and analyzed by classical bacteriological method (culture) and / or real-time PCR.

For mothers, the collection of 3-5 ml of milk when breastfeeding.

Monitoring schedule:

Day 21 and day 60 post delivery:

the following samples for search of GBS for will be performed to gather the primary endpoint:

For the mother:

* Vaginal sample.
* Collection of 3-5 ml of breast milk when breastfeeding

For the newborn:

* Sample collection of feces
* Swab of buccal cavity

Processing bacteriological samples:

All samples will be subjected to bacteriological analysis and DNA extraction for detection of GBS. GBS isolated will be identified and stored at - 80 ° C in a declared biological collection. DNA extracts will also stored at -20 ° C in a declared biological collection. All samples for microbiological analysis will be stored at - 80 ° C.

ELIGIBILITY:
Inclusion Criteria:

* Patient having a positive vaginal swab for GBS at the end of pregnancy (PCR +).
* Patient aged over 18 years
* Patient who received information and agreeing to sign informed consent
* Patient affiliated or beneficiary of an insurance

Exclusion Criteria:

- Patient does not speak and does not understand French

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 949 (Actual)
Dates: Start 2012-11-12 (Actual); Primary Completion 2015-06-03 (Actual); Study Completion 2015-06-03 (Actual)

PRIMARY OUTCOMES:
Detection of the hyper-virulent ST17 clone of Group B Strep | at 60 days post delivery
  Detection of the hyper-virulent ST17 clone of Group B Strep (GBS) in the prevention of neonatal GBS meningitis. The main objective is to demonstrate that the hypervirulent ST17 GBS clone colonizing the mother and postpartum acquired colonizes and persists at 60 days post delivery in the gut of new born significantly more than non-ST17 GBS strains.

SECONDARY OUTCOMES:
Digestive colonization | at day 21
  Digestive colonization of ST17 clone of Group B Strep in the newborns
Milk colonization | at day 21 and day 60
  Colonization of milk by ST17 clone of Group B Strep
Vaginal colonization | at day 21 and day 60
  Vaginal colonization by ST17 clone of Group B Strep
Late neonatal infections | between 3 weeks and 60 days
  Late neonatal infections will be observed between 3 weeks and 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Claire POYART, MD, PhD, Principal Investigator — Cochin Hospital
Locations (2):
- France (2):
  - Louis Mourier Hospital, Colombes
  - Cochin Hospital, Paris

REFERENCES:
- [Background] Tazi A, Plainvert C, Anselem O, Ballon M, Marcou V, Seco A, El Alaoui F, Joubrel C, El Helali N, Falloukh E, Frigo A, Raymond J, Trieu-Cuot P, Branger C, Le Monnier A, Azria E, Ancel PY, Jarreau PH, Mandelbrot L, Goffinet F, Poyart C. Risk Factors for Infant Colonization by Hypervirulent CC17 Group B Streptococcus: Toward the Understanding of Late-onset Disease. Clin Infect Dis. 2019 Oct 30;69(10):1740-1748. doi: 10.1093/cid/ciz033. PMID 30946447
- [Background] Plainvert C, El Alaoui F, Tazi A, Joubrel C, Anselem O, Ballon M, Frigo A, Branger C, Mandelbrot L, Goffinet F, Poyart C. Intrapartum group B Streptococcus screening in the labor ward by Xpert(R) GBS real-time PCR. Eur J Clin Microbiol Infect Dis. 2018 Feb;37(2):265-270. doi: 10.1007/s10096-017-3125-2. Epub 2017 Oct 29. PMID 29082442